CLINICAL TRIAL: NCT07115121
Title: Comparison of the Mean Change in Hemoglobin With Ferric Carboxymaltose and IV Iron Sucrose in Anemic Antenatal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Shamsa-BVH
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric Carboxymaltose-Group (Experimental): Patients were given ferric carboxymaltose as a maximum single dose of 1000 mg diluted in 250 mL of sterile 0.9% normal saline as a slow infusion over 45 minutes.
  Interventions: Drug: Intravenous Ferric Carboxymaltose
- Iron Sucrose-Group (Experimental): Patients received intravenous injections of iron sucrose complex, which contained 200 mg of elemental iron (equivalent to 2 ampoules of 5 ml), mixed in 100 ml of 0.9% normal saline and infused over a period of 30 minutes every other day for up to 5 doses.
  Interventions: Drug: Intravenous Iron Sucrose

INTERVENTIONS:
Drug: Intravenous Ferric Carboxymaltose — Patients were given ferric carboxymaltose as a maximum single dose of 1000 mg diluted in 250 mL of sterile 0.9% normal saline as a slow infusion over 45 minutes.
  Arms: Ferric Carboxymaltose-Group
Drug: Intravenous Iron Sucrose — Patients received intravenous injections of iron sucrose complex, which contained 200 mg of elemental iron (equivalent to 2 ampoules of 5 ml), mixed in 100 ml of 0.9% normal saline and infused over a period of 30 minutes every other day for up to 5 doses.
  Arms: Iron Sucrose-Group

SUMMARY:
Literature search has shows that both ferric carboxymaltose and iron sucrose complex are equally effective. Unfortunately, local data addressing this issue is scarce. To get further local data, the current study was planned with the objective to compare the mean change in hemoglobin with ferric carboxymaltose and IV iron sources in anemic antenatal patients in our local population.

DETAILED DESCRIPTION:
It was hypothesized that there was a difference in mean change in hemoglobin with ferric carboxymaltose as compared to IV iron sources in anemic antenatal patients. The findings of the study would be a valuable addition to the existing stats, and if the hypothesis stands correct, a large number of women of reproductive age would benefit from effective iron replacement therapy, with a comparatively low incidence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Aged 18 to 40 years
* Presented with anemia
* Any parity
* Gestational age < 12 weeks on LMP

Exclusion Criteria:

* Females with a history of hypertension
* Type II diabetes mellitus
* Gestational diabetes mellitus
* Ischemic heart disease
* Endocrine disorder
* Hematological disorders (hemophilia, leukemia, lymphoma, or myeloma)
* History of taking iron-lowering drugs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Increase in hemoglobin | 12 weeks
  Baseline hemoglobin was subtracted from post-treatment hemoglobin to assess increase in the hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be share on a reasonable request.